CLINICAL TRIAL: NCT05943509
Title: Feasibility of a Hearing Program in Primary Care for Underserved Older Adults
Brief Title: Hearing Program in Primary Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-00648
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Deafness
MeSH Terms: conditions — Deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alternative Rehabilitation Strategies (Experimental): Patients who screened positive for hearing loss and were randomized into the counselling on alternative rehabilitation strategies intervention arm.
  Interventions: Behavioral: Alternative rehabilitation strategies
- Usual Care (Active Comparator): Patients who screened positive for hearing loss and were randomized into the usual care audiology pathway control arm alone.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Alternative rehabilitation strategies — Counseling intervention.
  Arms: Alternative Rehabilitation Strategies
Behavioral: Usual Care — Usual care audiology pathway.
  Arms: Usual Care

SUMMARY:
During a primary care visit, investigators will screen and identify participants with hearing loss and then randomize to a) counseling on accessible assistive listening devices or b) referral to traditional audiology care pathway alone.

ELIGIBILITY:
Inclusion Criteria:

* speaks English or Spanish;
* capacity to consent to research

Exclusion Criteria:

• has or uses hearing aids or cochlear implants

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of Potential Participants Approached | Up to Month 3
Number of Potential Participants Screened | Up to Month 3
Percentage of Screened Participants with Hearing Loss | Up to Month 3

SECONDARY OUTCOMES:
Percentage of Intervention Arm Participants who Complete Counseling Session | Up to Month 3
Percentage of Participants who Respond to Outreach to Confirm Recommendations within 72 Hours | Up to Month 3
Percentage of Participants who Respond to 3-Month Follow-Up | Month 3

CONTACTS AND LOCATIONS:
Overall Officials: David Friedmann, Principal Investigator — NYU Langone Health
Locations (1):
- NYC H+H/Bellevue, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: David.friedmann@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to David.friedmann@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT05943509/ICF_000.pdf